CLINICAL TRIAL: NCT05838066
Title: A Randomized, Controlled, Open-label, Multicenter, Phase Ш Clinical Study of the Efficacy and Safety of KN026 in Combination With HB1801 Versus Trastuzumab in Combination With Pertuzumab and Docetaxel in the First-line Treatment of Subjects With HER2-positive Recurrent or Metastatic Breast Cancer.
Brief Title: Efficacy and Safety of KN026 in Combination With HB1801 in the First-line Treatment of Subjects With HER2-positive Recurrent or Metastatic Breast Cancer.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KN026-003
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: First-line Treatment of HER2-positive Recurrent or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Trastuzumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KN026+HB1801 (Experimental): Subjects will receive an intravenous (IV) infusion of KN026 plus HB1801. All subjects are required to receive study treatment as planned until investigator-assessed loss of benefit, toxic intolerance, withdrawal of consent, loss to follow-up, or death, whichever occurrs first.
  Interventions: Drug: Recombinant Humanized Bispecific antibody against HER2，KN026; Drug: HB1801
- Trastuzumab + Pertuzumab + Docetaxel (Active Comparator): On Day 1 of each 21-day cycle, patients will receive an intravenous (IV) infusion of Pertuzumab 840 mg loading dose followed by 420 mg per cycle, IV, D1, Q3W, in combination with trastuzumab 8 mg/kg loading dose followed by 6 mg/kg per cycle, IV, D1, Q3W and docetaxel 75 mg/m^2. All subjects are required to receive study treatment as planned until investigator-assessed loss of benefit, toxic intolerance, withdrawal of consent, loss to follow-up, or death, whichever occurred first.
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: Docetaxel

INTERVENTIONS:
Drug: Recombinant Humanized Bispecific antibody against HER2，KN026 — IV infusion
  Arms: KN026+HB1801
Drug: HB1801 — IV infusion
  Arms: KN026+HB1801
Drug: Pertuzumab — 840 mg loading dose followed by 420 mg per cycle, D1 Q3W, IV infusion
  Arms: Trastuzumab + Pertuzumab + Docetaxel
Drug: Trastuzumab — 8 mg/kg loading dose followed by 6 mg/kg per cycle, D1 Q3W, IV infusion
  Arms: Trastuzumab + Pertuzumab + Docetaxel
Drug: Docetaxel — 75 mg/m^2, D1 Q3W, IV infusion
  Arms: Trastuzumab + Pertuzumab + Docetaxel

SUMMARY:
This is a randomized, controlled, open-label, multicenter, phase Ш clinical study designed to compare the efficacy and safety of KN026 in combination with HB1801 to trastuzumab in combination with pertuzumab and docetaxel in the first-line treatment of subjects with HER2-positive recurrent or metastatic breast cancer. The statistical assumption for this study is superiority. The primary study endpoint was PFS as assessed by Blinded Independ Review Committee (BIRC).

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy and safety of KN026 combined with HB1801 versus trastuzumab combined with pertuzumab and docetaxel as first-line treatment for HER2-positive recurrent or metastatic breast cancer. This study will establish an independent data monitoring committee (IDMC) to conduct safety assessments after approximately 20 subjects in the treatment group complete the first cycle of treatment. During the safety assessment period, the study will continue to enroll subjects, and safety review meetings will be at 1 year of randomization in the first subject. In addition, the IDMC plans to conduct one interim analysis of efficacy during the study period.

The primary study hypotheses are that the combination of KN026 combined with HB1801 is superior to trastuzumab combined with pertuzumab and docetaxel with respect to: Progression-free Survival (PFS) as assessed by the BIRC per Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

ELIGIBILITY:
Key Inclusion Criteria:

* Voluntarily enrolled in this study and signed an informed consent form (ICF).
* Age ≥ 18 years.
* Recurrent or metastatic breast cancer confirmed by histology and/or cytology.
* Latest tumor tissue sample confirmed as HER2 positive by central laboratory testing.
* No prior systemic chemotherapy and/or HER2-targeted therapy for recurrent or metastatic breast cancer.
* Eastern Cooperative Oncology Group (ECOG) physical status score of 0 - 1.
* Presence of lesion (RECIST 1.1).
* Adequate organ and bone marrow function

Key Exclusion Criteria:

* Ineligible for any of the agents on the study
* Untreated or unstable parenchymal metastases, spinal cord metastases or compression, or carcinomatous encephalitis.
* Pregnant or lactating women.
* Presence of other circumstances that may interfere with the subject's participation in the study procedures or are inconsistent with the maximum benefit of the subject's participation in the study or affect the results of the study: e.g., history of mental illness, drug or substance abuse, any other disease or condition of clinical significance, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2023-07-23 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Free-progression survival (PFS) as evaluated by BIRC (RECIST1.1). | Up to approximately 4 years

SECONDARY OUTCOMES:
PFS (investigator assessment, RECIST1.1) | Up to approximately 4 years
Overall survival (OS) | Up to approximately 4 years
Objective response rate (ORR) | Up to approximately 4 years
Disease control rate (DCR) | Up to approximately 4 years
Duration of response (DoR) | Up to approximately 4 years
Frequency and severity of TEAE and SAE | Up to approximately 4 years
Concentration of KN026 in serum | Up to approximately 4 years
Concentration of HB1801 in serum | Up to approximately 4 years
Incidence of KN026 Anti-drug antibody (ADA) and neutralizing antibody (Nab) (if applicable) | Up to approximately 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials Information Group, Beijing, chaoyang, China

IPD SHARING:
Plan to Share IPD: No